CLINICAL TRIAL: NCT04943796
Title: Prevalence of ADHD and Health Outcomes in Adult Outpatients With Psychiatric Disorders: a Multi-country, Two-part, Observational Study
Brief Title: A Study to Learn About the Occurrence of ADHD in Adults With Mental Conditions and Their Quality of Life
Acronym: LANDSCAPE
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-489-4004; MACS-2020-070101 (Other: Takeda)
Record Dates: First submitted 2021-06-28; First posted 2021-06-29 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Part I: Participants with ADHD: Participants with psychiatric disorders undergoing ADHD diagnosis.
- Part II: Participants with ADHD: To collect pseudonymized data from participants who are underdiagnosed of ADHD with psychiatric disorders in daily clinical practice for up to 9 months from both Part I and II.

SUMMARY:
The main aim of the study is to find out how frequently adults with at least one psychiatric condition have ADHD (but have not been diagnosed with ADHD before) and to describe the quality of life of these adults who have been diagnosed with ADHD. To find out how often ADHD is not diagnosed in these adults could provide awareness about this condition and could help to improve preventing underdiagnosis.

ELIGIBILITY:
Inclusion criteria:

Part I:

* Adult greater than or equal to (>=)18 years of age or Canadian adult >=19 years of age
* Ability to consent, as judged by the study investigator
* Diagnosis of at least one psychiatric disorder of at least 12 months duration, based on International classification of diseases (ICD)-10 codes registered in electronic health records
* Consecutive assessment for ADHD (as per routine clinical practice)
* Able to read and write in the first language of the respective country

Part II

* Inclusion in study Part I
* Diagnosis of ADHD during Part I, according to routine diagnostic procedure and algorithms
* Anticipated availability for being followed over 9 months

Exclusion criteria:

Part I:

* Diagnosis of any of the following at any time prior to signing informed consent: schizoaffective disorder, intellectual disability, or other cognitive disorders
* Occurrence of any of the following events within the 6 months prior to signing consent: psychotic episodes, acute intoxication, or psychotropic drug withdrawal syndrome.
* Diagnosis of ADHD at any time before study inclusion
* Serious and unstable medical condition (severe disease that limits survival to 1 year)
* Participation in a clinical interventional trial in the 12 months prior signing consent

Part II:

- Participant being followed-up for ADHD in a different site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with diagnosis of any of the following psychiatric disorder: Major depressive disorder (MDD), Anxiety disorders (AD), Bipolar disorders (BD), Substance use disorders (SUD), Border line disorder and Binge eating disorder.
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Part I: Percentage of Participants With Positive or Negative ADHD Diagnosis | At baseline
  Percentage of participants with positive or negative ADHD diagnosis will be reported.
Part II: Change From Baseline in Quality of Life- questionnaire (AAQoL) by Overall Psychological/Psychiatric Clinical Management | Baseline, 3 Month and 9-Month of follow-up
  AAQoL (32) is an instrument designed to evaluate the quality of life in ADHD adult participants It has 29 items organized in four domains: Life Productivity (11 items); Psychological Health (6 items), Life Outlook (7 items) and Relationships (5 items). Each item is rated with a five-point Likert scale ranging from 1= Not at all/Never to 5=Extremely/Very Often. Total and domain-specific scores are computed by reversing scores for all items, except those in the Life Outlook domain; transforming all item scores to a 0 to100 point scale (1=0; 2=25; 3=50; 4=75; 5=100); and summing the item scores and dividing by them by item count. Total score ranges from 0 to 100 with higher score representing better quality of life. Change from baseline in AAQoL by overall psychological/psychiatric clinical management will be reported.
Part II: Change From Baseline in AAQoL by ADHD-Specific Clinical Management | Baseline, 3-month, and 9-month follow up
  AAQoL (32) is an instrument designed to evaluate the quality of life in ADHD adult participants It has 29 items organized in four domains: Life Productivity (11 items); Psychological Health (6 items), Life Outlook (7 items) and Relationships (5 items). Each item is rated with a five-point Likert scale ranging from 1= Not at all/Never to 5=Extremely/Very Often. Total and domain-specific scores are computed by reversing scores for all items, except those in the Life Outlook domain; transforming all item scores to a 0 to100 point scale (1=0; 2=25; 3=50; 4=75; 5=100); and summing the item scores and dividing by them by item count. Total score ranges from 0 to 100 with higher score representing better quality of life. Change from baseline in AAQoL by ADHD-Specific Clinical Management will be reported.

SECONDARY OUTCOMES:
Part I: Percentage of Participants With Confirmed Diagnosis of ADHD Based on Adult ADHD Self-Reporting Scale (ASRS) | At baseline
  ASRS is designed to evaluate for severity of symptoms as specified in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). ASRS is composed of 18 questions, and uses a scale that ranges from 0-4 based on the individuals mark in either the "never, rarely, sometimes, often, very often" column for a possible total score of 72. The minimum score to qualify for study inclusion is 8 (i.e. 4 or more "symptom-positive" answers), and the maximum possible score is 72. The higher the score, the more indicative of higher severity of ADHD symptoms. Each column is used to describe the severity of the individuals symptoms based on the questions asked. Each participant is asked to make a mark within one column for each question that best describes their answer. Percentage of participants with confirmed diagnosis of ADHD in participants with psychiatric disorder based on adult ASRS will be reported.
Part I: Percentage of Participants With Confirmed Diagnosis of ADHD Based on Diagnostic Interview for Adult ADHD (DIVA 5.0) | At baseline
  DIVA 5.0 is a structured diagnostic interview for Adult ADHD, and is based on the criteria for ADHD in DSM-5. Whenever possible the DIVA should be completed with adults in the presence of a partner and/or family member, to enable retrospective and collateral information to be ascertained at the same time. The DIVA usually takes around one and a half hours to complete. The DIVA only asks about the core symptoms of ADHD required to make the DSM-IV diagnosis of ADHD, and does not ask about other co-occurring psychiatric symptoms, syndromes or disorders. In this study, participant will be interviewed using DIVA only if scores in ASRS showed positive diagnosis of ADHD.
  Percentage of participants with confirmed diagnosis of ADHD in participants with psychiatric disorder based on DIVA 5.0 will be reported.
Part I: Percentage of Participants With Confirmed Diagnosis of ADHD Based on Diagnostic and Statistical Manual of Mental Disorders (DSM-5) | At baseline
  DSM-5 confirm the diagnosis of ADHD if meeting all of the following criteria: (i) having five out of nine ADHD inattention and/or hyperactivity/impulsivity symptoms for the last 6 months or more; (ii) having several symptoms before the 12 years of age; (iii) having several symptoms in at least two settings (e.g., at home or work; and with friends or family members); (iv) having symptoms interfering with quality of social, academic, or occupational functioning; and (v) having symptoms that do not occur exclusively during the course of a psychotic disorder and are not better explained by another mental disorder.
  Percentage of participants with confirmed diagnosis of ADHD in participants with psychiatric disorder based on DSM-5 will be reported.
Part II: Number of Modalities for Non-ADHD Psychiatric/Psychological clinical management | Baseline, 3 Month and 9-Month of follow-up
  Number of modalities for non-ADHD psychiatric/psychological clinical management will be assessed.
Part II: Type of Treatment Given to Participants with ADHD for Non-ADHD Psychiatric/Psychological Clinical Management | Baseline, 3 Month and 9-Month of follow-up
  Type of treatment given to participants with ADHD for non-ADHD psychiatric/psychological clinical management will be assessed.
Part II: Duration of Treatment for Non-ADHD Psychiatric/Psychological Clinical Management | Baseline, 3 Month and 9-Month of follow-up
  Duration of treatment for non-ADHD psychiatric/psychological clinical management will be assessed.
Part II: Number of Modalities for ADHD-specific Psychiatric/Psychological Clinical Management | Baseline, 3 Month and 9-Month of follow-up
  Number of modalities for ADHD-specific psychiatric/psychological clinical management will be assessed.
Part II: Type of Treatment Given to Participants with ADHD for ADHD-Specific Overall Psychiatric/Psychological Clinical Management | Baseline, 3 Month and 9-Month of follow-up
  Type of treatment given to participants with ADHD for ADHD-specific overall psychiatric/psychological clinical management will be assessed.
Part II: Duration of Treatment for ADHD-Specific Psychiatric/Psychological Clinical Management | Baseline, 3 Month and 9-Month of follow-up
  Duration of treatment for ADHD-specific psychiatric/psychological clinical management will be assessed.
Part II: Change From Baseline in Functional Assessment Short Test (FAST) Score | Baseline, 3 Month and 9-Month of follow-up
  FAST is a brief instrument designed to assess the main functioning problems experienced by psychiatric participants, particularly bipolar participants. It comprises 24 items that assess impairment or disability in six specific areas of functioning: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time. The scale used to evaluate functionality is the FAST Scale, the minimum value being 0 and maximum value of 72, domain scores are scaled in a negative direction (i.e. lower scores denote higher functionality).
Part II: Change From Baseline in Clinical Global Impressions Scale- Severity of Illness (CGI-S) | Baseline, 3 Month and 9-Month of follow-up
  CGI-S is a 7-point scale to rate the participant's severity of illness at the time of assessment, relative to the clinician's past experience with participants who have the same diagnosis by means of one question: Considering your total clinical experience with this particular population, how mentally ill is the participant at this time which is rated on the following seven-point scale with range from 1 to 7 were: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill participants.
Part II: Change From Baseline in Clinical Global Impressions Scale- Improvement (CGI-I) Score | Baseline, 3 Month and 9-Month of follow-up
  CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention: Compared to the participant's condition at admission to the project [prior to medication initiation], this participant's condition ranges from 1 to 7 were: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.
Change From Baseline in Health Resource Utilization (HRU) | Baseline, 3 Month and 9-Month of follow-up
  Utilization of health resources by the study population during the 12 months prior ADHD assessment in the total sample and according to the diagnosis will be assessed at baseline, 3-months and 9 months follow up.
Part II: Functionality Level and Quality of Life by ADHD-Specific Clinical Management | Baseline, 3-month, and 9-month follow up
  Continues variables (e.g., age, functionality scores, quality of life scores, number of previous visits to the hospital) and categorical variables (e.g., sex, clinical characteristics, psychiatric disorders, ADHD warning signs, treatments, previous tests) will be described in the total sample and according to confirmed/no confirmed ADHD; and will be compared using T-test or ANOVA test (continues variables) and Chi squared test (categorical variables).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (14):
- Canada (3):
  - Pacific Coast Recovery Care, Burnaby, British Columbia
  - Hopital de Psychiatrie de Trois-Rivières, Pavillon St-Joseph, Trois-Rivières, Quebec
  - Regina Mental Wellness Clinic, Regina, Saskatchewan
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinik und Poliklinik für Psychiatrie und Psychoterapie, Bonn
  - Universitätsklinikum Frankfurt am Main, Frankfurt am Main
  - Asklepios Klinikum Hamburg, Hamburg
- Spain (3):
  - Hospital Vall d'Hebron, Barcelona
  - Clínica Dr. Quintero, Madrid
  - Hs. Infanta Elena, Madrid
- Psykiatrisk klinik Umeå, Umeå, Sweden
- University Hospitals of Geneva, Geneva, Switzerland
- United Kingdom (2):
  - Cumbria Northumb, Tyne & Wear FT, Adult Psychiatry Dept, Newcastle upon Tyne
  - Tees Esk and Wear Valley foundation, York

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60dc8cc1ef0b71001e743dfc